CLINICAL TRIAL: NCT01779648
Title: The Influence of the Different Ways of Pneumatic Compression on Clinical and Physiologic Efficacies in Preventing Deep Vein Thrombosis: a Randomised Comparative Study
Brief Title: Comparison of Different Intermittent Pneumatic Compression Devices for Deep Vein Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: DS MAREF Co., Ltd. (Unknown); Small and Medium Business Administration, KOREA (Unknown)
Responsible Party: Principal Investigator, Jae-Sung Choi, Associate Professior, Thoracic and Cardiovascular Department, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPCDVT
Record Dates: First submitted 2013-01-27; First posted 2013-01-30 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Venous Thrombosis; Deep Vein Thrombosis
Keywords: deep vein thrombosis; intermittent pneumatic compression; venous hemodynamics
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simultaneous compression+Fixed refill time (Active Comparator): Simultaneous bilateral compression with fixed venous refill time through the whole duration of pneumatic compression
  Interventions: Device: DVT-3000
- Alternate compression+Adjusted refill time (Active Comparator): alternate bilateral compression with adjusted venous refill time which would change several times during pneumatic compression
  Interventions: Device: SCD Express

INTERVENTIONS:
Device: DVT-3000
  Other Names: Simultaneous sequential intermittent pneumatic compression; Fixed venous refill time
  Arms: Simultaneous compression+Fixed refill time
Device: SCD Express
  Other Names: Alternate and sequential intermittent pneumatic comression; Adjusted venous refill time
  Arms: Alternate compression+Adjusted refill time

SUMMARY:
Various kinds of intermittent pneumatic compression devices (IPC) with particular ways of compression have been developed and used for prevention of deep vein thrombosis.

There are still some controversies about the physiologic properties and clinical impact of numerous issues including the variety of the cuff length, inflation rate, compression sequence, compression-relaxation cycle rate, and pressure generation characteristics.

This study is designed to compare clinical efficacies as well as venous hemodynamic improvements between Simultaneous bilateral compression with fixed venous refill time versus alternate compression with adjusted refill time

ELIGIBILITY:
Inclusion Criteria:

* the patients who undergo total knee replacement arthroplasty

Exclusion Criteria:

* (1) chronic superficial or deep venous insufficiency, (2) venous anomalies like duplication of the superficial femoral vein, (3) previous venous thromboembolism history, (4) being under anticoagulation therapy, (5) severe arteriosclerosis obliterans without palpable dorsalis pedis pulse, (6) open fracture, hemorrhagic condition, or extensive dermatitis at lower legs, (7) congestive heart failure. Additional exclusion criteria included a documented malignant tumor, because pharmacologic prophylaxis with anticoagulants would be more reasonable in this case.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Sung Choi, Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started in March, 2012 and ended in January, 2013. A total 57 participants were recruited and tested for enrollment after admission to the hospital.
Pre-assignment Details: Two of them were excluded prior to group assignment because of the detection of a lung cancer and a deep vein thrombosis, respectively.
Groups:
- Group SF: Simultaneous bilateral compression with fixed venous refill time through the whole duration of pneumatic compression
  Simultaneous compression +Fixed refill time:
- Group AA: alternate bilateral compression with adjusted venous refill time which would change several times during pneumatic compression
  Alternate compression+Adjusted refill time
Period: Overall Study
Arm/Group | Group SF | Group AA
Started | 28 | 27
Completed | 27 | 27
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group SF: Simultaneous bilateral compression with fixed venous refill time through the whole duration of pneumatic compression
  simultaneous compression :
- Group AA: alternate bilateral compression with adjusted venous refill time which would change several times during pneumatic compression
  alternate compression :
- Total: Total of all reporting groups
Arm/Group | Group SF | Group AA | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 9
  >=65 years | 20 | 26 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.1) | 72.3 (5.9) | 70.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 28 | 27 | 55
Body Mass Index [Mean (Standard Deviation); unit: kg/m2]
  Female | 27.1 (5.2) | 26.3 (4.4) | 26.7 (4.8)
  Male | 26.5 (4.6) | 28.0 (1.6) | 27.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Deep Vein Thrombosis
Description: Computed tomographic angiography were performed on 4th postoperative days to detect deep vein thrombosis and evaluate its extent and location.
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Population: One participant of Group SF dropped out of the analysis due to the device error; air leakage in the closed circuit system.
Measure: Number; unit: participants
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
participants
  Deep vein thrombosis | 14 | 15
  ipsilateral development | 9 | 12
  contralateral development | 1 | 1
  bilateral development | 4 | 2
  distal DVT | 13 | 14
  proximal DVT | 1 | 1
  Symptomatic DVT | 0 | 0
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p = 0.785, Chi-squared

2. Secondary Outcome: Peak Velocity
Description: Doppler ultrasonography were performed to measure one of the venous hemodynamic parameters to be compared. A longitudinal scans of bilateral superficial femoral veins, just distal to the confluence of the profunda femoral veins, were performed. Baseline velocity, flow pattern, and augmented flow of 11 seconds (Simultaneous compression arm) or 12 seconds (Alternate compression arm) were recorded. Under fixed state of other ultrasound scan parameters, peak velocity (PV) was measured by determination of maximum point of the augmented waveform.
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
cm/sec | 24.8 (5.9) | 22.8 (4.9)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Mean of right and left leg values were compared between the two device groups; Test type: Superiority or Other; p = 0.195, t-test, 2 sided

3. Secondary Outcome: Mean Velocity
Description: Doppler ultrasonography were performed to measure one of the venous hemodynamic parameters to be compared. A longitudinal scans of bilateral superficial femoral veins, just distal to the confluence of the profunda femoral veins, were performed. Baseline velocity, flow pattern, and augmented flow of 11 seconds (Alternate compression arm) or 12 seconds (Simultaneous compression arm) were recorded. This is an automatically measured mean value of venous flow.
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
cm/sec | 10.0 (2.5) | 9.7 (2.7)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Mean of right and left leg values were compared between the two device groups; Test type: Superiority or Other; p = 0.722, t-test, 2 sided

4. Secondary Outcome: Peak Volume Flow
Description: Doppler ultrasonography were performed to measure one of the venous hemodynamic parameters to be compared. A longitudinal scans of bilateral superficial femoral veins, just distal to the confluence of the profunda femoral veins, were performed. Baseline velocity, flow pattern, and augmented flow of 11 seconds (Simultaneous compression arm) or 12 seconds (Alternate compression arm) were recorded. Peak volume flow (PVF) was automatically calculated with 1-second interval around the PV.
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
mL/min | 205.3 (76.5) | 176.4 (72.1)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Mean of right and left leg values were compared between the two device groups; Test type: Superiority or Other; p = 0.158, t-test, 2 sided

5. Secondary Outcome: Total Volume Flow
Description: Doppler ultrasonography were performed to measure one of the venous hemodynamic parameters to be compared. A longitudinal scans of bilateral superficial femoral veins, just distal to the confluence of the profunda femoral veins, were performed. Baseline velocity, flow pattern, and augmented flow of 11 seconds (Simultaneous compression arm) or 12 seconds (Alternate compression arm) were recorded. Total volume flow (TVF) was automatically calculated by the software.
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
mL/min | 160.9 (58.1) | 144.2 (59.0)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Mean of right and left leg values were compared between the two device groups; Test type: Superiority or Other; p = 0.301, t-test, 2 sided

6. Secondary Outcome: Expelled Total Volume
Description: Expelled volume was theoretically calculated value in order to figure out how much blood was squeezed by the compression for an hour; expelled total volume (ETV) = single cycle augmented TVF x cycling rate (cycles/hour).
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/hour
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
mL/hour
  right leg | 7214.0 (3389.2) | 4342.0 (2419.0)
  left leg | 6102.8 (3957.6) | 3334.5 (1390.5)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Age, sex, body mass index, and baseline TVF (total volume flow) are controlled as fixed-effects parameters

7. Secondary Outcome: Expelled Peak Volume
Description: Expelled volume was theoretically calculated value in order to figure out how much blood was squeezed by the compression for an hour; expelled peak volume (EPV) = single cycle augmented PVF x cycling rate (cycles/hour).
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/hour
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
mL/hour
  right leg | 999.8 (344.3) | 633.1 (321.4)
  left leg | 904.0 (454.2) | 525.5 (196.2)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Age, sex, body mass index, and baseline PVF (peak volume flow) are controlled as fixed-effects parameters

8. Secondary Outcome: Augmented PV
Description: Enhanced peak velocity by application of intermittent pneumatic compression
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
cm/sec
  right | 62.8 (17.8) | 56.2 (19.5)
  left | 57.1 (20.2) | 58.5 (18.8)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis; Age, sex, body mass index, and baseline PV (peak velocity)are controlled as fixed-effects parameters

9. Secondary Outcome: Augmented MV
Description: Enhanced mean velocity by application of pneumatic compression
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
cm/sec
  right leg | 20.4 (9.6) | 18.2 (4.7)
  left leg | 33.1 (6.1) | 18.3 (6.1)

10. Secondary Outcome: Augmented PVF
Description: Enhanced peak volume flow by application of pneumatic compression
Time Frame: On 4th postoperative days after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/min
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
mL/min
  right leg | 666.5 (229.5) | 514.6 (465.0)
  left leg | 602.7 (302.8) | 465.0 (186.6)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Age, sex, body mass index, and baseline peak volume flow are controlled as fixed-effects parameters

11. Secondary Outcome: Augmented TVF
Description: Enhanced total volume flow by application of pneumatic compression
Time Frame: on 4th postoperative day after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: mL/min
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
mL/min
  right leg | 400.7 (188.2) | 324.2 (150.5)
  left leg | 339.0 (219.8) | 271.2 (135.8)
Statistical Analysis 1: Comparison: Group SF vs Group AA; Test type: Superiority or Other; p = 0.132, Mixed Models Analysis; Age, sex, body mass index, and baseline total volume flow are controlled as fixed-effects parameters

12. Secondary Outcome: Cycling Rate
Description: Number of cuff inflation-deflation cycle during an hour. In group SF, the cycling rate is fixed as 90 cycles/hour, but in group AA, it is variable according to the individual venous refill time.
Time Frame: on 4th postoperative day after total knee replacement arthroplasty
Measure: Mean (Standard Deviation); unit: cycles/hour
Units Other Than Participants: limbs
Arm/Group | Group SF | Group AA
Number analyzed (Participants) | 27 | 27
Number analyzed (limbs) | 54 | 54
cycles/hour | 90 (0) | 78.9 (20.4)

ADVERSE EVENTS:
Arm/Group | Group SF | Group AA
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 6/27 | 5/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group SF (N=27) | Group AA (N=27)
operative wound oozing (Musculoskeletal and connective tissue disorders) | 1 | 1
wound pain aggravation (Musculoskeletal and connective tissue disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes